CLINICAL TRIAL: NCT04192617
Title: A Randomized,Placebo Controlled, Double-blind, Parallel Group, Phase II Study to Evaluate the Efficacy and Safety of SM03, Compared to Placebo, in Patients With Moderate-to-Severe Active Rheumatoid Arthritis Receiving Methotrexate
Brief Title: A Study to Evaluate the Safety and Efficacy of SM03 in Patients With Rheumatoid Arthritis Receiving Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SinoMab BioScience Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM03-RA-II-V3.3
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SM03 600 mg*2 (Experimental): SM03: 600 mg intravenous (IV) on week 0,2, and week 12,14; placebo: 600 mg intravenous (IV) on week 4 and16; Methotrexate: 7.5-20 mg/wk oral.
  Interventions: Drug: SM03; Drug: Placebo; Drug: Methotrexate
- SM03 600 mg*3 (Experimental): SM03: 600 mg intravenous (IV) on week 0,2, 4, and week 12,14,16; Methotrexate: 7.5-20 mg/wk oral.
  Interventions: Drug: SM03; Drug: Methotrexate
- placebo*3 (Placebo Comparator): placebo: 600 mg intravenous (IV) on week 0,2, 4, and week 12,14,16; Methotrexate: 7.5-20 mg/wk oral.
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: SM03 — SM03: 600 mg intravenous (IV)
  Arms: SM03 600 mg*2; SM03 600 mg*3
Drug: Placebo — Placebo: 600 mg intravenous (IV)
  Arms: SM03 600 mg*2; placebo*3
Drug: Methotrexate — methotrexate: 7.5-20 mg/week oral

SUMMARY:
This study evaluated the safety and efficacy of SM03 compared to placebo in patients with active rheumatoid arthritis(RA) receiving methotrexate

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-75 years of age.
* Rheumatoid arthritis (RA) for ≥ 12 months, diagnosed according to the revised 1987 American College of Rheumatology (ACR) criteria for the classification of rheumatoid arthritis.
* Moderate to severe active RA with swollen joint count (SJC) ≥ 8 (66 joint count), and tender joint count (TJC) ≥ 8 (68 joint count) at screening and baseline.
* At screening, either C-reactive protein (CRP) ≥ 0.6 mg/dL (6 mg/L), or Erythrocyte sedimentation rate (ESR) ≥ 28 mm/hour, or Morning stiffness of joint for ≥ 45 minutes
* Inadequate response to methotrexate, having received and tolerated at a dose of 7.5-20 mg/week for ≥ 12 weeks, at a stable dose over the past 4 weeks.

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA.
* Use of any biological DMARDs for RA within past 6 months.
* Concurrent treatment with any Disease Modifying Anti-Rheumatic Drug (DMARD) other than methotrexate
* Active infection, or history of serious or chronic infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2016-02-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 24 | Week 24
  To achieve an ACR20 required at least a 20% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 20% improvement in three of the following five additional measurements:
  * Physician's global assessment of disease activity (assessed using a 10 cm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (assessed using a 10 cm VAS);
  * Patient's assessment of pain (assessed using a 10 cm VAS);
  * Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3);
  * Acute phase reactant: C-reactive protein (CRP)

SECONDARY OUTCOMES:
Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 4,8,12, 16 | Week 4,8,12,16
  To achieve an ACR20 required at least a 20% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 20% improvement in three of the following five additional measurements:
  * Physician's global assessment of disease activity (assessed using a 10 cm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (assessed using a 10 cm VAS);
  * Patient's assessment of pain (assessed using a 10 cm VAS);
  * Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3);
  * Acute phase reactant: C-reactive protein (CRP)
Percentage of Participants With an ACR50 Response at Week 24 | Week 24
  To achieve an ACR50 required at least a 50% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 50% improvement in three of the following five additional measurements:
  * Physician's global assessment of disease activity (assessed using a 10 cm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (assessed using a 10 cm VAS);
  * Patient's assessment of pain (assessed using a 10 cm VAS);
  * Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3);
  * Acute phase reactant: C-reactive protein (CRP)
Percentage of Participants With an ACR70 Response at Week 24 | Week 24
  To achieve an ACR70 required at least a 70% improvement compared with Baseline in both tender joint counts (68 joints assessed for tenderness) and swollen joint counts (66 joints assessed for swelling), as well as a 70% improvement in three of the following five additional measurements:
  * Physician's global assessment of disease activity (assessed using a 10 cm Visual Analog Scale [VAS]);
  * Patient's global assessment of disease activity (assessed using a 10 cm VAS);
  * Patient's assessment of pain (assessed using a 10 cm VAS);
  * Health Assessment Questionnaire (HAQ; a patient completed questionnaire consisting of 20 questions, scored from 0-3);
  * Acute phase reactant: C-reactive protein (CRP)
Change From Baseline in Disease Activity Score (DAS28-ESR) at Week 24 | Baseline and Week 24
  The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * Erythrocyte sedimentation rate (ESR);
  * Patient's global assessment of disease activity measured on a 10 cm visual analog scale.
  The DAS28 score ranges from zero to ten. A DAS28 score above 5.1 means high disease activity whereas a DAS28 less than or equal to 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6.
Percentage of Participants With European League Against Rheumatism (EULAR) Response at Week 24 | Week 24
  A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS28 score. The DAS28 score ranges from 0-10, with higher scores indicating more disease activity.
  A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score of less than or equal to 3.2.
  A Moderate Response is defined as either:
  an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 from Baseline and attainment of a DAS28 score of less than or equal to 5.1 or, an improvement (decrease) in the DAS28 of more than 1.2 from Baseline and attainment of a DAS28 score of greater than 3.2.
  No Response is defined as either an improvement (decrease) in the DAS28 of less than or equal to 0.6, or an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 of more than 5.1.
Percentage of Participants With Adverse Events | Week 0 to 24
  Percentage of participants who reported an AE or SAE, a drug-related AE, who had an acute infusion reaction, an AE leading to study drug discontinuation, with an infection or serious infection, or who died.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hostipal, Beijing, China

REFERENCES:
- [Derived] Li J, Li M, Wu D, Zhou J, Leung SO, Zhang F. SM03, an anti-human CD22 monoclonal antibody, for active rheumatoid arthritis: a phase II, randomized, double-blind, placebo-controlled study. Rheumatology (Oxford). 2022 May 5;61(5):1841-1848. doi: 10.1093/rheumatology/keab699. PMID 34508557